CLINICAL TRIAL: NCT03394053
Title: Investigating the Mechanistic Biology of Primary Immunodeficiency Disorders
Brief Title: The Mechanistic Biology of Primary Immunodeficiency Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180041; 18-I-0041
Record Dates: First submitted 2018-01-05; First posted 2018-01-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-16

CONDITIONS: Primary Immunodeficiency Disorders
Keywords: SCID; Natural Killer (NK) cell deficiency; Combined Immunodeficiency; T-Cell Lymphocytopenia; Of Immune Pathways; Natural History
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected Patient: Person with a clinical diagnosis of a PID (age 0-90); either known or unknown as defined by lab and/or clinical findings on 2 or more occasions that are consistent with a defect in innate or adaptive immunity
- Normal Volunteer: Persons (age 18-75 years) who are not related to another study subject, who do not have a PID, weight >110lbs, no history of viral hepatitis B or C, have a negative HIV screening test
- Relative of Patient: Biological relatives (age 0-90 years) of a subject who meets affected patient criteria, but who do not have a PID themselves

SUMMARY:
Background:

Primary immunodeficiency disorders, or PIDs, are diseases that weaken the immune system. This makes it easier for a person to get sick. Some PIDs are mild and may not be diagnosed until later in life. Other kinds are severe and can be identified shortly after birth. Researchers want to learn more about PIDs by comparing data from relatives and healthy volunteers to people with a PID.

Objective:

To learn more about PIDs, including their genetic causes.

Eligibility:

People ages 0-90 with a PID or their healthy biological relatives the same ages

Healthy volunteers ages 18-75

Design:

Participants will be screened with a medical history, physical exam, and HIV blood test. They may have a pregnancy test.

Participants may repeat the screening tests.

Blood taken at screening will be used for genetic tests and research tests. Participants will be told test results that affect their health. Some blood will be stored for future research.

Adult participants with a PID may have a small piece of skin removed. The area will be numbed. A small tool will take a piece of skin about the size of a pencil eraser.

Researchers may collect fluid or tissue samples from PID participants regular medical care. They will use them for research tests.

Participants with a PID will have 3 follow-up visits over 10 years (for infants, 2 years). Visits will include a physical exam, medical history, and blood draw.

Participants with a PID and their relatives will be called once a year for 10 years. They will talk about how they are feeling and if they have developed any new symptoms or illnesses.

...

DETAILED DESCRIPTION:
This is a natural history study designed to investigate forms of primary immunodeficiency disorders (PIDs), and to better define both new and previously described forms of PID, including severe combined immunodeficiency (SCID), combined immunodeficiency, natural killer (NK) cell deficiency, and other disorders. Patients with clinical and/or laboratory evidence of PID will be recruited at Children s National Health System (CNHS) and the National Institute of Allergy and Infectious Diseases (NIAID). Infants identified at birth with a positive newborn screening for SCID and confirmed to have T-cell lymphocytopenia will also be recruited at CNHS. Subjects with a known or unknown PID and infants with T-cell lymphocytopenia will provide one or more blood samples during the course of the study to enable immunologic and genetic investigations of immune pathways contributing to PIDs. These subjects will also be followed clinically to longitudinally assess the natural history of novel and known PIDs. Subjects will be followed over time with regard to their immunologic phenotype, clinical disease (including incidence of infections, autoimmune phenomena, allergic disease, or malignancies), and response to both preventative and definitive therapies. Biological relatives who do not have PID and healthy adult volunteers will also be eligible to serve as controls for this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects must meet one of the following 4 criteria:

     1. Patients (age 0-90 years) with a clinical diagnosis of a form of PID (either known or unknown). PID is defined by laboratory and/or clinical findings on two or more occasions that are consistent with a defect in innate or adaptive immunity. Specific PIDs are defined by the International Union of Immunological Societies guidelines. These subjects must also be willing to undergo genetic testing and to allow their biospecimens to be modified into iPS cells. Women of childbearing potential, or who are pregnant or lactating, may be eligible. The volume of blood collected for research purposes will be reduced, and no skin biopsies will be performed for research purposes in consideration of their safety.
     2. Infants identified at birth with positive newborn screening for SCID and confirmed to have T-cell lymphocytopenia. These subjects must be willing to undergo genetic testing.
     3. Biological relatives (age 0-90 years) of a subject who meets criterion 1a or 1b but who do not have a PID themselves. All relatives must be willing to undergo genetic testing. Women of childbearing potential, or who are pregnant or lactating, may be eligible. The volume of blood collected for research purposes will be reduced in consideration of their safety.
     4. Healthy volunteers (age 18-75 years) who are not related to another study subject, who do not have a PID, whose weight is greater than 110 pounds, do not have a history of any heart, lung, or kidney disease, or bleeding disorders, do not have a history of viral hepatitis (B or C), and have a negative HIV screening test.
  2. All subjects must be willing to allow their samples to be stored for future research.

EXCLUSION CRITERIA:

1. Subjects with secondary causes of immunodeficiency are excluded from this study. Secondary causes of immunodeficiency include HIV infection and immunodeficiency that is deemed to be secondary to chronic use of immunosuppressive medications or chemotherapeutic agents.
2. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential subjects with confirmed or suspected PID and their biological relatives will be referred to the study from physicians at CNHS or at the NIH. In addition, patients who have a clinical diagnosis of PID may also be referred from physicians at other institutions. Healthy volunteers may be recruited from the NIH Clinical Research Volunteer Program
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of unique clinical phenotypes associated with known genetic causes of PID. | 10- 15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Identification of genetic variants that are associated with PID. | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.

SECONDARY OUTCOMES:
Overall survival | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Incidence of malignancies. | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Incidence of infections. | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Incidence of autoimmune disease | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Incidence of allergic disorders | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Impact of both preventative and definitive treatments on event-free survival (as defined by survival in absence of invasive or chronic infection, autoimmunity, or malignancies). | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.
Identification of phenotypic, molecular, and functional abnormalities associated with known or novel forms of PID. | 10-15 years
  comparing these subjects to the large cohort of data in the Exome Aggregation Consortium (ExAC) Browser (Beta), which is available through http://exact.broadinstitute.org.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi D Notarangelo, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - Children's National Health System (CNHS), Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-I-0041.html